CLINICAL TRIAL: NCT06298318
Title: Effect of Acute Binge Drink Intervention on Healthy Young Subjects: a Double-blinded, Randomized Trial
Brief Title: Metabolic Changes in Healthy Subjects with Acute Binge Drink
Acronym: MeABD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Li Lab,MD, Professor, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Acute Binge Drink; NSFC: 82273625 (Other Grant/Funding Number: National Natural Science Foundation of China); ZCLY24H2602 (Other Grant/Funding Number: Natural Science Foundation of Zhejiang Province); 202410344043 (Other Grant/Funding Number: National Project for Innovation and Entrepreneurship Training Program for College Students); 202410344075X (Other Grant/Funding Number: National Project for Innovation and Entrepreneurship Training Program for College Students)
Record Dates: First submitted 2023-11-01; First posted 2024-03-07 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Binge Drinking; Liver Injury; Hepatic Steatosis
Keywords: Acute alcohol intake; Liver
MeSH Terms: conditions — Binge Drinking; Fatty Liver | interventions — Water

STUDY DESIGN:
Intervention Model Description: not involve drug or biologic products
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): BMI: if 18.5 ≤ BMI < 24.0, individuals received 1.0 g/kg body weight of water; if 24.0 ≤ BMI ≤ 28.0, individuals received 0.8 g/kg body weight of water.
  Interventions: Other: water
- vodka group (Experimental): BMI: if 18.5 ≤ BMI < 24.0, individuals received 1.0 g/kg body weight of vodka; if 24.0 ≤ BMI ≤ 28.0, individuals received 0.8 g/kg body weight of vodka.
  Interventions: Other: Vodka

INTERVENTIONS:
Other: Vodka — BMI: if 18.5 ≤ BMI < 24.0, individuals received 1.0 g/kg body weight of vodka; if 24.0 ≤ BMI ≤ 28.0, individuals received 0.8 g/kg body weight of vodka.
  Arms: vodka group
Other: water — equal amount of non-alcoholic beverages with the same taste and colour but without alcohol
  Arms: Control group

SUMMARY:
The goal of this double-blinded, randomized trial is to investigate the effects of acute binge drinking on liver function, liver fat content, and lipid metabolism in healthy young subjects. The main questions it aims to answer are:

1. If acute binge drinking could alleviate liver injury and hepatic steatosis.

DETAILED DESCRIPTION:
The goal of this double-blinded, randomized trial is to investigate the effects of acute binge drinking on liver function, liver fat content, and lipid metabolism in healthy young subjects. The main questions it aims to answer are:

1. If acute binge drinking could alleviate liver injury and hepatic steatosis.

Participants will be randomized into two groups (n=40) and provided vodka (1 g/kg body weight) or an equal amount of non-alcoholic beverages with the same taste and colour but without alcohol, respectively. 15 minutes later, they are successively provided with the same breakfast. Venous blood samples were collected at 0h, 1h, 3h, 5h, 6h, 12h, and 24h from each subject, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. male aged 18-30 years;
2. body mass index (BMI) ranging from 18.5 to 28 kg/m²;
3. having prior experience with binge drinking or hangovers, as assessed using the Personal Assessment of Maximum Drinking Capacity Survey Questionnaire

Exclusion criteria

1. with alcohol intolerance or alcohol dependence;
2. with serious health conditions, such as liver, kidney, cardiovascular, or gastrointestinal diseases;
3. vegetarians;
4. smokers;
5. with a history of drug use, including antihistamines, antihypertensives, antidiabetics, anxiolytics, and central nervous system depressants;
6. who had used antibiotics within two weeks prior to the trial;
7. who had consumed alcohol, alcoholic beverages or alcohol-containing foods within one week before the trial.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-27 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
hepatic function change | day1-2 of each 0 hour and 1hour and 5hours and 12 hours and 24 hours
  Research blood hepatic function include:Alanine Aminotransferase in U/L;Aspartate Aminotransferase in U/L;Gamma-Glutamyltransferase in U/L;Alpha-Fucosidase in U/L;Alkaline Phosphatase in U/L;cholinesterase in U/L;Lactate Dehydrogenase Enzyme in U/LTBIL in μmol/L, direct bilirubin in μmol/L, indirect bilirubin in μmol/L, and total bile acid in μmol/L
Hepatic fibrosis change | day1-2 of each 0 hour and 1hour and 5 hours and 12 hours and 24 hours
  Research blood hepatic fibrosis include:Hyaluronicacid in ng/mL;Laminin in ng/mL;type # in ng/mL;precollagen in ng/ mL;type # collagen in ng/mL;Fibronect in ng/mL
Lipid metabolism change | day1-2 and of each 0 hour and 1hour and 5 hours and 12 hours and 24 hours
  Research blood Fat metabolism include:Triglycerides in mmol/L;HDL-Cholesterol in mmol/L;LDL--Cholesterol in mmol/ L;Apolipoprotein A in mmol/L;Apolipoprotein B in mmol/L;Lipoprotein(a) in mmol/L

SECONDARY OUTCOMES:
Ethanol concentration | day1-2 of each 0 hour and 1hour and 5hours and 12 hours and 24 hours
  Ethanol concentration change in mg/dL of each set
Acetaldehyde concentration | day1-2 of each 0 hour and 1hour and 5hours and 12 hours and 24 hours
  Acetaldehyde concentration change in mg/dL of each set

OTHER OUTCOMES:
Fecal metabolites | day1-2 of each 0 hour and 24 hours
  Gut microbial communities and their abundant features will be analysed based on shotgun metagenomic sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: guiiqin sun, Study Chair — Zhejiang Chinese Medical University
Locations (1):
- Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Protect volunteers' personal health data and personal privacy

REFERENCES:
- [Background] Lee MH, Kwak JH, Jeon G, Lee JW, Seo JH, Lee HS, Lee JH. Red ginseng relieves the effects of alcohol consumption and hangover symptoms in healthy men: a randomized crossover study. Food Funct. 2014 Mar;5(3):528-34. doi: 10.1039/c3fo60481k. PMID 24458173
- [Background] Kim H, Kim YJ, Jeong HY, Kim JY, Choi EK, Chae SW, Kwon O. A standardized extract of the fruit of Hovenia dulcis alleviated alcohol-induced hangover in healthy subjects with heterozygous ALDH2: A randomized, controlled, crossover trial. J Ethnopharmacol. 2017 Sep 14;209:167-174. doi: 10.1016/j.jep.2017.07.028. Epub 2017 Jul 24. PMID 28750942